CLINICAL TRIAL: NCT06615817
Title: Comparison Between 14/10 Intermittent Fasting and the Southern Italian Mediterranean Diet in the Variation of NAFLD Score, Inflammatory Indices and Intestinal Microbiota
Brief Title: Intermittent Fasting, Mediterranean Diet and NAFLD
Acronym: RC2024-21
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis (Other)
Responsible Party: Principal Investigator, Dr. Rosa Reddavide - MSc, Principal Investigator, Biologyst, Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC2024-21
Record Dates: First submitted 2024-09-18; First posted 2024-09-27 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: NAFLD; Obesity; Intermittent Fasting; Mediterranean Diet
Keywords: Obesity; Liver Diseases
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity; Intermittent Fasting; Liver Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group - Mediterranean diet with low glycemic index (No Intervention): Control group in which patients will follow a Mediterranean diet with a low glycemic index
- Case group - Intermittent Fasting (Experimental): Intermittent fasting 14/10 with 14 hours of nocturnal fasting and 10 hours of feeding with a low glycemic index Mediterranean diet.
  Interventions: Dietary Supplement: Intermittent Fasting

INTERVENTIONS:
Dietary Supplement: Intermittent Fasting — In this group, a diet based on intermittent fasting will be administered - with 14 hours of nocturnal fasting and 10 hours of feeding with a low glycemic index Mediterranean diet.
  Arms: Case group - Intermittent Fasting

SUMMARY:
This study aims to evaluate the effects of Intermittent Fasting (IF) 14/10 compared with the Low Glycemic Index Mediterranean Diet on NAFLD.

DETAILED DESCRIPTION:
Interventional, randomized, controlled 2-arm clinical trial

The two study arms are:

* Low-Glycemic Index Mediterranean Diet (Control Arm).
* IF 14/10 (Experimental Arm) with 14 hours of overnight fasting and 10 hours of feeding with Low Glycemic Index Mediterranean Diet.

The study involves the enrollment of 60 subjects (30 in each arm) with NAFLD, medium/severe grade diagnosed by Fibroscan, randomly assigned using randomization tables to one of the two study arms.

The duration of the nutritional intervention is 4 months. During the study duration period, patients will undergo 3 visits.

At T0 (Screening Visit) patients, who are potentially enrollable, after signing the informed consent, will undergo:

* Medical history (family, physiological, remote and upcoming pathological and pharmacological);
* Fibroscan, to assess the degree of hepatic steatosis;
* Survey of anthropometric characteristics (BMI, abdominal circumference, neck circumference);
* Bioimpedance examination;
* NuWell (Nutrition Wellness Survey) questionnaire completion.
* IPAQ (Daily Physical Activity Questionnaire) questionnaire.

In case the inclusion criteria are met, the enrolled patients will be randomized, using randomization tables, into one of the two arms under the study.

The enrolled patients, will be invited to return after 7 days to complete T0 and receive the personalized food plan, depending on the arm they belong to and anthropometric characteristics.

Fasting for at least 12 hours, they will undergo blood sampling by venipuncture and body composition assessment by DEXA.

Enrolled subjects will be asked to bring a stool sample and a urine sample for fecal and urinary mycriobiota and metabolome analysis.

Patients will be given the Food Diary, which must be reported completed at each visit.

After 2 months from the start of treatment (T0 + 60gg) patients will be called for T1.

At this visit, patients who have been fasting for at least 12 hours will undergo:

* Samples by venous puncture;
* Bioimpedance examination;
* Anthropometric measurements. Patients will be asked to bring a stool sample and a urine sample, and the Food Diary will be checked.

After another 2 months (T1 + 60gg: End of treatment) patients will be called for T2.

At this visit, patients, fasting for at least 12 hours, will undergo:

* Samples by venous puncture;
* Fibroscan
* Bioimpedance examination;
* DEXA
* Anthropometric measurements. Patients will be asked to bring a stool sample and a urine sample, and a Food Diary will be collected.

The blood sample taken will be used to assay routine hematochemical parameters and nutritional, metabolic and cardiovascular risk. Specifically, the following will be assayed: blood glucose, glycated hemoglobin, insulin, azotemia, creatinine, total cholesterol, LDL cholesterol, HDL cholesterol, triglycerides, urate, AST, ALT, gamma GT, total protein, protein electrophoresis, high-sensitivity PCR, TSH, FT3, FT4, blood count, ferritin, vitamin D, prolactin, cortisol, urine tests, IL 1, 4, 6, 8, 10, CK18 and TNFα.

Patients will be given the reports of Routine blood tests only, Fibroscan, Bioimpedance Examination and DEXA.

ELIGIBILITY:
Inclusion Criteria:

* Medium/severe NAFLD (CAP>268)
* BMI between 25 and 35

Exclusion Criteria:

* diabetes treated with insulin,
* fatty liver disease linked to alcohol consumption,
* chronic inflammatory intestinal and oncological diseases,
* visceral obesity which does not allow good resolution of Fibroscan images,
* subjects in serious medical conditions that may compromise participation in the trial,
* people following a special diet or unable to follow a diet for religious or other reasons.
* Pregnancy and breastfeeding

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
The effect of intervention on CAP value | at Baseline and after 4 months
  To evaluate the change in hepatic steatosis score after 4 months of a low glycemic index Mediterranean diet and 14/10 intermittent fasting with a low glycemic index Mediterranean diet.
  The cut off to indicate the presence of steatosis is CAP>268. A decrease in the CAP value indicates an improvement in the pathology

SECONDARY OUTCOMES:
The effect of the intervention on the Body Composition detected with DEXA | at Baseline and after 4 months
  Evaluate the change in body composition detected with DEXA after 4 months of a low glycemic index Mediterranean diet and 14/10 intermittent fasting with a low glycemic index Mediterranean diet
The effect of the intervention on the Body Composition detected with bioimpedance analysis | at Baseline and after 4 months
  Evaluate the change in body composition detected with bioimpedance analysis after 4 months of a low glycemic index Mediterranean diet and 14/10 intermittent fasting with a low glycemic index Mediterranean diet

OTHER OUTCOMES:
The effect of intervention on routine blood chemistry parameters, relating to NAFLD | at Baseline and after 4 months
  To evaluate whether a low glycemic index Mediterranean diet and 14/10 intermittent fasting with a low glycemic index Mediterranean diet can exert favorable effects on the parameters of routine blood tests relating to NAFLD,after 4 months.
  The regression formula for prediction of NAFLD is based on 6 variables: age (years), BMI(kg/m2), IFG/diabetes, AST/ALT ratio, platelet count and albumin (g/dl).
The effect of intervention on routine blood chemistry parameters, relating to fibrosis | at Baseline and after 4 months
  To evaluate whether a low glycemic index Mediterranean diet and 14/10 intermittent fasting with a low glycemic index Mediterranean diet can exert favorable effects on the parameters of routine blood tests relating to fibrosisafter 4 months.
  We will take into consideration the FIB4 value. The formula for FIB-4 is: Age ([yr] x AST [U/L]) / ((PLT [10(9)/L]) x (ALT [U/L])(1/2)).
The effect of intervention on routine blood chemistry parameters, relating to nutritional status | at Baseline and after 4 months
  To evaluate whether a low glycemic index Mediterranean diet and 14/10 intermittent fasting with a low glycemic index Mediterranean diet can exert favorable effects on the parameters of routine blood tests relating to nutritional status, after 4 months.

REFERENCES:
- [Background] Zelber-Sagi S, Godos J, Salomone F. Lifestyle changes for the treatment of nonalcoholic fatty liver disease: a review of observational studies and intervention trials. Therap Adv Gastroenterol. 2016 May;9(3):392-407. doi: 10.1177/1756283X16638830. Epub 2016 Mar 17. PMID 27134667
- [Background] Laferrere B, Panda S. Calorie and Time Restriction in Weight Loss. N Engl J Med. 2022 Apr 21;386(16):1572-1573. doi: 10.1056/NEJMe2202821. No abstract available. PMID 35443112
- [Background] Marinac CR, Nelson SH, Breen CI, Hartman SJ, Natarajan L, Pierce JP, Flatt SW, Sears DD, Patterson RE. Prolonged Nightly Fasting and Breast Cancer Prognosis. JAMA Oncol. 2016 Aug 1;2(8):1049-55. doi: 10.1001/jamaoncol.2016.0164. PMID 27032109